CLINICAL TRIAL: NCT01074502
Title: An Open-label, Single-arm Pilot Study of the Safety and Efficacy of an Oral PDE4-inhibitor Agent, Apremilast, in the Treatment of Moderate to Severe Acne
Brief Title: Apremilast in the Treatment of Moderate to Severe Acne
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding due to Celgene administrative decision
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Aida Lugo-Somolinos, MD, Associate Professor of dermatology, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CELG0001
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-02

CONDITIONS: Acne
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- apremilast (Experimental): apremilast 20 mgs twice a day for 12 weeks
  Interventions: Drug: apremilast

INTERVENTIONS:
Drug: apremilast — apremilast 20 mgs orally twice a day for 12 weeks

SUMMARY:
Acne is a chronic inflammatory disease of the pilosebaceous unit that affects 80-90% of the population, especially teenagers, although adult acne is a significant problem for 3-6 % of adult men and 5-12% of adult women. Although acne is not a life-threatening disease, it produces significant psychological disturbances and permanent skin scars.

A novel anti-inflammatory, not antibiotic drug may be an excellent alternative for the treatment of moderate to severe acne. Apremilast has been shown to inhibit the production of tumor necrosis factor (TNF)-alpha, IL-8 and neutrophil infiltration, all of which are elevated in inflammatory acne.

Our intention is to study Apremilast in the treatment of moderate to severe acne.

DETAILED DESCRIPTION:
The hypothesized sequence of events in inflammatory acne starts with the formation of a microcomedone with accumulation of cornified keratinocytes within the follicle. Presence and/or proliferation of P.acnes induces the production of IL-1 alpha, tumor necrosis factor (TNF)- alpha, IL-8 and granulocyte-macrophage colony-stimulating factor (GM-CSF). Inflammation caused by CD4+ T cells causes a T-helper 1 cytokine response mediated by Toll-like receptors (TLR)-2 and TLR-4 whose expression is increased by P. acnes. Infiltration by neutrophils appears 72 hrs after, with possible disruption of the follicular wall and more inflammation. TNF-alpha liberated by keratinocytes stimulates the activation of pro-matrix metalloproteinase (MMP)-2 activity in the dermis with remodeling by fibroblasts with the consequence of possible scarring.

The usual treatment for moderate to severe inflammatory acne involves the use of long-term topical retinoids and antibiotics such as doxycycline or minocycline that had been showed to decrease the inflammatory response as well as decreasing the population of P. acnes. Since acne is a long term condition, several years of antibiotics are usually required. Recently, the problematic of antibiotic overuse has received great attention and concerns. Chronic antibiotic use has been implicated in increasing the risk of breast cancer and upper respiratory infections, and there is also a concern for antibiotic resistance. Recent recommendations by the Global Alliance to Improve Outcomes in Acne Group include the limitation for the use of oral antibiotics to a maximum of 3 months. So there is a need to find alternatives that does not include the use of oral antibiotics.

The only effective and available treatment for severe acne is isotretinoin which may have potential serious side effects. Lately also it has been implicated in the development of depression and suicidal ideations in the teenager population.

A novel anti-inflammatory, not antibiotic drug may be an excellent alternative for the treatment of moderate to severe acne. Apremilast has been shown to inhibit the production of tumor necrosis factor (TNF)-alpha, IL-8 and neutrophil infiltration, all of which are elevated in inflammatory acne. Preliminary data of the use of Apremilast in psoriasis makes us believe that this medication is safe for short-term use in acne patients.

Our intention is to study Apremilast in the treatment of moderate to severe acne.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Must be male or female and aged 18-45 years of age, inclusive, at time of consent and be in general good health.
* Must be able to adhere to the study visit schedule and other protocol requirements
* Moderate to severe acne ( a 3 or 4 score in the RGA) of the face at Baseline.
* Subjects with 17-100 non-inflammatory lesions (open and closed comedones) and with 25-150 inflammatory lesions (papules and pustules) and 0-15 nodules (no larger than 1 cm each) and no cystic lesions.
* Must meet the following laboratory criteria:

  * Hemoglobin > 12 g/dL
  * White blood cell (WBC) count ≥ 3000 /mL (≥ 3.0 X 109/L) and ≤ 14,000/mL (< 14 X 109/L)
  * Platelets ≥ 100,000 /mL (≥ 100 X 109/L)
  * Serum creatinine ≤ 1.5 mg/dL (or ≤ 133 μmol/L)
  * Total bilirubin < 2.0 mg/dL
  * Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]) < 1.5x upper limit of normal (ULN)

    * Negative ANA
    * Negative cANCA
    * Negative antiphospholipid antibodies
* Females of childbearing potential (FCBP)‡ must have a negative urine pregnancy test at screening (Visit 1). In addition, sexually active FCBP must agree to use TWO of the following adequate forms of contraception while on study medication: oral, injectable, or implantable hormonal contraceptives; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner while on study. A FCBP must agree to have pregnancy tests every 4 weeks while on study medication.
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with FCBP while on study medication and for 84 days after taking the last dose of study medication
* If a moisturizer or sunscreen is needed during the study, subjects must be willing to accept only acceptable products (non-comedogenic and without ingredients that may worsen or improve acne such as Cetaphil cleanser and Neutrogena oil-free moisturizer).

Exclusion Criteria:

* Inability to provide voluntary consent
* Use of any topical acne treatment (salicylic acid, benzoyl peroxide, retinol, antibiotics) 2 weeks prior to Baseline.
* Use of topical astringents or antimicrobial soaps for one week prior to Baseline.
* Use of any topical retinoid, systemic antibiotic or topical or systemic corticosteroids in the face 4 weeks prior to Baseline.
* Use of a systemic retinoid, such as isotretinoin, 6 months prior to Baseline
* Any confluent nodule, cyst and/or sinus tract present.
* Any nodule larger than 10 mm.
* Subjects who are using medications that can exacerbate acne such as mega-doses of vitamin D, vitamin B2, B6, B12, haloperidol, halogens such as iodide and bromide, lithium, hydantoin and Phenobarbital). Multivitamins, iron supplements and folate are acceptable, but should be used consistently throughout the study.
* Subjects who have had a facial procedure (chemical or laser peel, blue light treatment, microdermabrasion, etc) within 4 weeks before enrollment or during the study.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Subjects who abuse drugs or alcohol (drug screening not required).
* Pregnant, trying to become pregnant or breastfeeding.
* Use of estrogens, androgens or hormonal contraception or devices for less than 12 weeks prior to Baseline. Subjects are allowed to enroll as long as they do not expect to change dose, product, or discontinue use during the study.
* Systemic fungal infection
* History of active mycobacterial infection with any species (including Mycobacterium tuberculosis) within 3 years prior to screening visit. Subjects with Mycobacterium tuberculosis infection more than 3 years prior to screening visit are allowed if successful treatment was completed at least 3 years prior to randomization and is documented and available for verification.
* Mycobacterium tuberculosis infection as indicated by a positive Purified Protein Derivative [PPD] skin test (>15mm induration). Subjects with a positive PPD skin test are ineligible.
* History of incompletely treated Mycobacterium tuberculosis infection as indicated by

  * Subject's medical records documenting incomplete treatment for Mycobacterium tuberculosis
  * Subject's self-reported history of incomplete treatment for Mycobacterium tuberculosis
* History of recurrent bacterial infection (at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years)
* Clinically significant abnormality on the chest x-ray (CXR) at screening. Chest x-rays performed within 3 months prior to start of study drug are acceptable.
* Use of any investigational medication within 4 weeks prior to start of study drug or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer)
* Any clinically significant abnormality on 12-lead ECG at screening
* History of congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency [CVID])
* Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening
* History of Human Immunodeficiency Virus (HIV) infection
* Antibodies to Hepatitis C at screening
* Malignancy or history of malignancy (except for treated [ie, cured] basal-cell skin carcinomas > 3 years prior to screening )

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aida Lugo-Somolinos, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University Of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apremilast
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Apremilast
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Success Rate (Based on the Researcher's Global Assessment (RGA) Sum of Clear (0) or Almost Clear (1))
Description: RGA measures the severity of acne. The scale goes from 0-4. 0 will be better and 4 will be worse. Scores can only be whole numbers (0,1,2,3,4)ordinal.
Time Frame: Baseline to 16 weeks
Population: small number of subjects to analyze
Arm/Group | Apremilast
Number analyzed (Participants) | 0

2. Primary Outcome: Percentage of Patients With a Minimum 2-grade Improvement in the Researcher Global Assessment (RGA) From Baseline to Week 12.
Description: RGA measures the severity of acne. The scale goes from 0 (better)to 4 (worse). Score can only be whole numbers, ordinal.
Time Frame: Baseline to 12 weeks
Population: small number of subjects to be analyzed
Arm/Group | Apremilast
Number analyzed (Participants) | 0

3. Primary Outcome: Mean Percentage Change From Baseline in Individual Lesion Counts (Total, Inflammatory, Non-inflammatory) at Week 12
Time Frame: Baseline to 12 weeks
Arm/Group | Apremilast
Number analyzed (Participants) | 0

4. Secondary Outcome: The Absolute Change in Lesion Counts (Total, Inflammatory, Non-inflammatory) From Baseline to Week 12
Time Frame: Baseline to12 weeks
Arm/Group | Apremilast
Number analyzed (Participants) | 0

5. Secondary Outcome: Safety of Apremilast 20 Mgs BID for 12 Weeks Will be Assessed by Evaluating Adverse Events (AEs), Vital Signs, Laboratory Evaluations and Withdrawals From the Study
Description: Number of participants with adverse events
Time Frame: Baseline to 16 weeks
Arm/Group | Apremilast
Number analyzed (Participants) | 0

6. Primary Outcome: Percentage of Patients Achieving a Clear or Almost Clear PGA at 16 Weeks
Time Frame: Baseline to 16 weeks
Arm/Group | Apremilast
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Apremilast
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes